CLINICAL TRIAL: NCT00540566
Title: Optical Biopsy of Human Skin in Conjunction With Laser Treatment
Status: Completed | Type: Observational
Sponsor: University of California, Irvine (Other)
Collaborators: Beckman Laser Institute University of California Irvine (Other)
Responsible Party: Principal Investigator, Beckman Laser Institute and Medical Center, J.S.Nelson, MD,PhD,Professor of Surgery and Biomedical Engineering, University of California, Irvine
Other Study IDs: 1996200
Record Dates: First submitted 2007-10-04; First posted 2007-10-08 (Estimated); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: Malignant Melanoma; Merkel Cell Carcinoma; Basal Cell Carcinoma; Squamous Cell Carcinoma; Atypical Nevi; Congenital Nevi; Seborrheic Keratosis; Paget's Disease; Dermatofibroma; Kaposi's Sarcoma; Port Wine Stain; Hemangioma; Tattoos; Scleroderma; Burns
MeSH Terms: conditions — Melanoma; Carcinoma, Merkel Cell; Carcinoma, Basal Cell; Carcinoma, Squamous Cell; Dysplastic Nevus Syndrome; Keratosis, Seborrheic; Osteitis Deformans; Histiocytoma, Benign Fibrous; Sarcoma, Kaposi; Port-Wine Stain; Hemangioma; Scleroderma, Diffuse; Burns

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Optical Biopsy: Optical Biopsy imaging
  Interventions: Device: Optical Biopsy imaging

INTERVENTIONS:
Device: Optical Biopsy imaging — Optical Biopsy imaging

SUMMARY:
This study is to compare the ability of optical biopsy. Research can use light enters the skin, collected, analyzed by the computer, and a picture created for the pathologist to conventional histologic examination compare with the pathologist looking at the piece of tissue through a microscope makes the diagnosis.

DETAILED DESCRIPTION:
The Optical measurements provide quantitative optical property values that reflect changes in tissue perfusion, oxygen consumption, and cell/matrix development. Each measurement requires less than 5 minutes to execute. The measurements will be taken before and after skin treatment.This non-invasive, non-contact technique has great potential as a means to diagnose different skin problems without the need to obtain a piece of tissue from the skin.

ELIGIBILITY:
Inclusion Criteria:

* Male or female age > 18 years

Exclusion Criteria:

* current participation in any other investigational drug evaluation
* inability to understand and carry out instructions

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: primary care clinic, community sample
Sampling Method: Non-Probability Sample
Enrollment: 113 (Actual)
Dates: Start 1999-06; Primary Completion 2008-06 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
normal skin | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: John S Nelson, M.D,Ph.D, Principal Investigator — Beckman Laser Institue, University of California Irvine
Locations (1):
- Beckman Laser Institute, Unversity of California Irvine, Irvine, California, United States